CLINICAL TRIAL: NCT05592652
Title: Identification of the Clinical Specificities of Complex Posttraumatic Stress Disorder
Acronym: IDPLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220118-IDPLEX; 2022-A01206-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-10-13; First posted 2022-10-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: patients and volunteers will undergo a series of psychometric scales
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- simple post-traumatic stress disorder (Other): Patients suffering from PTSD according to DSM-5 diagnostic features
  Interventions: Other: Survey
- complex post-traumatic stress disorder (Other): Patients suffering from CPTSD according to CIM-11 diagnostic features
  Interventions: Other: Survey
- volonteer trauma + (Other): non clinical volunteer with traumatic exposure
  Interventions: Other: Survey
- volonteer trauma - (Other): non clinical volunteer without traumatic exposure
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey including demographic, clinical and psychopathological questions

SUMMARY:
Identification of the clinical specificities of complex post-traumatic stress disorder post-traumatic stress disorder

DETAILED DESCRIPTION:
In general, the current state of the literature in the field the lack of data on elements of characterization of PTSD compared to simple PTSD, which are which are essential for deciding on the discriminatory validity of discriminative validity of PTSD as a disorder in its own right disorder in its own right. The challenge of defining the nosographic scope of this disorder is twofold, since the links between diagnosis and treatment are decisive for developing treatments adapted to the treatments adapted to the psychopathology of the patients. These characterization elements are therefore crucial in order to improve the perspective of improving the effectiveness of future treatment which are currently lacking in TSPTC.

ELIGIBILITY:
Inclusion Criteria Patient :

* Age ≥ 18 years
* Free, informed and signed consent
* Affiliated to a social security scheme

Inclusion Criteria volonteer :

* Age ≥ 18 years
* Free, informed and signed consent
* Affiliated to a social security scheme

Exclusion Criteria (patient and volonteer):

* Under legal protection (curatorship, guardianship, safeguard of justice)
* Present a former or current psychotic disorder, a former or current neurological disease, a history of head trauma (loss of consciousness of more than 10 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Dissociation | baseline
  The Dissociation questionnaire (DIS-Q; Vanderlinden et al., 1993) is used to scan dissociative experience and disruptions, and to measure their severity. It can be used for psychiatric patients, individuals with traumatic experience, and for scanning purposes. Its instructions are available in the introduction section of the scale and patients are asked to mark the most appropriate option for their condition. It consists of a total of 63 questions and the subject marks one option for each of these questions. Each item is scored between 1 and 5 points, mean score is obtained by dividing total scores by 63. High scores reflect high dissociative experience and disruptions. This scale can distinguish the subjects with dissociative disorder from healthy individuals or from patients with schizophrenia or bipolar mood disorder.
Emotional dysregulation | 5 minutes for questionnaire completion
  The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) is a 36-item self-report questionnaire assessing emotion regulation difficulties. A typical item is "I am clear about my feelings". Items are rated from 1 (almost never) to 5 (almost always). The French version has good internal consistency for all the sub-dimensions, with Cronbach alpha values of 0.84 to 0.90 (Dan-Glauser & Scherer, 2013). The DERS provides a total score and higher values are associated with a stronger emotion regulation difficulties.
PTSD | baseline
  The Posttraumatic stress disorder Checklist Scale PCL-5 (Weathers et al., 2013) is a self-administered questionnaire to assess the severity of PTSD in the clinic and research according to DSM-5 criteria. This scale translated and validated in French (Ashbaugh et al., 2016) is composed of 20 items, rated from 1 (not at all) to 5 (very often) according to the intensity and frequency of symptoms in the past month. When adding the scores for each of the 20 items, a total score greater than or equal to 33 indicates probable PTSD. The PCL-5 has good psychometric qualities as it demonstrates strong internal consistency (α = .94) as well as good convergent (rs = .74 to .85) and divergent validity (rs = .31 to .60) (Blevins et al., 2015). This tool is also sensitive to therapeutic change and can be used in repeated measures as evidenced by strong test-retest reliability (r = .82) (Blevins et al., 2015).
Complex PTSD | baseline
  The International Trauma Questionnaire (ITQ; Cloitre et al., 2018) is a self-report measure of PTSD and CPTSD severity assessing the following symptoms : reeexperiencing, avoidance, sense of threat, affective dysregulation, negative self- concept and disturbances in relationships. Participants are asked to select on a Likert scale how much a symptom has been bothersome in the past month or how true certain statements are of them, with scores ranging from 0 ("not at all") to 4 ("extremely"). Diagnosis of PTSD requires the endorsement of one of two symptoms from each PTSD cluster, while CPTSD diagnosis requires the endorsement of one of two symptoms from both PTSD and 'Disturbances in Self-organization' clusters. Both diagnoses require the presence of functional impairment. The ITQ is the only validated measure for ICD-11 PTSD and CPTSD.

SECONDARY OUTCOMES:
Early Maladaptive Schema | 10 minutes for questionnaire completion
  The YSQ-S3 is a self-report measure assessing 18 early maladaptive schemas. The items are categorized in four schema factors which replaced Young's previous five schema domains (Young et al., 2003): Disconnection, Impaired Autonomy, Exaggerated Standards, and Impaired Limits (Hoffart, et al., 2005). Participants are asked to rate descriptive statements on a 6-step Likert-scale which ranges from "completely untrue of me" (1) to "describes me perfectly" (6). The YSQ-S3 provides a total score and higher values are associated with a stronger presence of early maladaptive schema. This measure has demonstrated good psychometric properties and has shown age neutrality when administered across the lifespan (Pauwels et al., 2014).
Personality Disorders | baseline
  The PDQ-4+ (Hyler, 1994) which includes 107 items, and which is used to evaluate 12 kinds of personality disorders in the DSM-IV system. The PDQ-4+ is a 99-item self-report measure of DSM-IV personality disorders on which items are answered using a yes/no format. Personality disorders symptom counts are computed by summing the yes items for each personality disorder. The PDQ-4+ provides a total score and higher values are associated with a stronger presence of personality disorders.
Depressive symptoms | baseline
  The PHQ-9 is used to assess depressive symptoms over the last two weeks (Kroenke et al., 2001). Respondents indicate on a 0-3 scale, the frequency with which they experience the following symptoms: (1) anhedonia, (2) depressed mood, (3) sleep disturbance, (4) fatigue, (5) appetite changes, (6) low self-esteem, (7) concentration problems, (8) psychomotor disturbances, and (9) suicidal ideation. Total scores range from 0 to 27, with scores ≥10 representing clinically significant depressive symptoms (Kroenke & Spitzer, 2002). Furthermore, the PHQ-9 is validated as a depressive symptom severity measure (total score 1-4: minimal depression, 5-9: mild depression, 10-14: moderate depression, 15-19: moderately severe depression, and 20-27: severe depression; Kroenke et al., 2001). The PHQ-9 demonstrates high internal consistency and good sensitivity and specificity for identifying cases of MDD (Kroenke et al., 2001).
Anxiety State and Trait | baseline
  The STAI consists for a 40 items self-evaluation questionnaire which includes separate measures of state and trait anxiety. The State-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how respondents' feel about anxiety "right now, at this moment" through four scales: one (not at all), two (somewhat), three (moderately so), and four (very much so). The Trait-anxiety scale consists of twenty statements that assess how people "generally feel" about anxiety with four scales: one (almost never), two (sometimes), three (often), and four (almost always). A rating of four indicates the presence of a high level anxiety and one indicates the absence of a high level anxiety (Spielberger et al., 1983). The anxiety level was found by calculation of scores, The range of scores is from 20-80, the higher the score indicating greater anxiety (Spielberger et al., 1983).
Peritraumatic Dissociation | Less than five minutes for questionnaire completion
  The Peritraumatic Dissociation Experiences Questionnaire (PDEQ) (Marmar et al., 1994) is a 10-item self-administered test measuring dissociative experiences during a traumatic event and in the minutes and hours following the event. Each item is scored from 1 (not at all true) to 5 (extremely true). A score of 15 or higher indicates significant peri-traumatic dissociation. The PDEQ has demonstrated good psychometric qualities in its original version (Marmar et al., 1994) and in its French version (Birmes et al., 2005). It has satisfactory test-retest reliability (r = .72) and internal consistency (α = .78), as well as good convergent validity with the PDI [15] and the IES-R (Brunet, St-Hilaire, Jehel & King, 2003, Birmes et al., 2005).
Peritraumatic Distress | baseline
  The Peritraumatic Distress Inventory (PDI) (Brunet et al., 2001) is a self-administered scale composed of 13 items. It measures the emotional distress reactions that a person experienced at the time of a traumatic event and in the minutes and hours following the event. These reactions are measured retrospectively from the DSM-4 PTSD criterion A. This scale identifies two factors; dysphoric emotions and perceived life threat. Each item is scored from 0 (not at all true) to 4 (extremely true). The total score is obtained by summing all items. A score of 15 or more indicates significant peri-traumatic distress.
Childhood Trauma | baseline
  The Childhood Trauma Questionnaire short-form (CTQ) is a standardized, retrospective 28-item self-report inventory that measures the severity of different types of childhood trauma (Bernstein & Fink, 1998). For each of the five clinical subscales, Emotional Abuse, Physical Abuse, Sexual Abuse, Emotional Neglect and Physical Neglect, the participants respond to each item in the context of "when you were growing up" and answer according to a five-point Likert scale ranging from "never" = 1 to "very often" = 5, producing scores of 5 to 25 for each trauma subscale. The higher the score the greater the severity of maltreatment. Scores above the recommended cut-off score for "low" severity on each of the subscales are considered cases of abuse and neglect (Bernstein & Fink, 1998).
Alcohol misuse | baseline
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item self-report instrument used for assessing alcohol misuse (Saunders, Aasland, Babor, de la Puente, & Grant, 1993). The measure contains two subscales assessing alcohol use (3 items; Cronbach's α = .85) and alcohol-related consequences (7 items; Cronbach's α = .83). Responses range from 0 to 40. Higher scores indicate greater likelihood of hazardous and harmful drinking. However, total scores of 8 or more are recommended as indicators of hazardous and harmful alcohol use, as well as possible alcohol dependence. As well, guidelines establish that AUDIT scores in the range of 8-15 represent a medium level of alcohol problems, scores in the range of 16-19 represent a high level of alcohol problems and scores of 20 or above clearly warrant further diagnostic evaluation for alcohol dependence. The validity and reliability of the AUDIT with early adult samples has been established (DeMartini & Carey, 2012).
Resilience | baseline
  Resilience will be measured using the French version of the Connor-Davidson Resilience Scale (CD-RISC; Connor & Davidson 2003). This 25-item self-administered questionnaire measures resilience by combining five factors (tenacity, sense of self-efficacy, emotional and cognitive control, adaptability, tolerance of negative affect). Each item is coded on a 5-point scale ranging from 0 to 4. The addition of the scores for each item gives an overall resilience score ranging from 0 to 100. The higher the score, the more resilient the individual. The CD-RISC-25 has demonstrated good psychometric qualities. A French version of the questionnaire has been validated.
Well Being | baseline
  The French version of the WHO-5 (World Health Organization-Five Well Being Index, 1999) was used to measure current mental well-being. It is a short, unidimensional, self-reported scale composed of 5 items ranged from 0 ("at no time") to 5 ("all the time"). Total score is obtained by adding all of the item scores. Total raw scores range from 0 to 25. High scores reflect a high well-being. The scale is known to have high psychometric and clinimetric properties (Topp et al., 2015) and used for both screening and clinical trial purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine TAPIA, PhD, Study Director — University of Bordeaux
Locations (1):
- UHTours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arntz A, Jacob GA, Lee CW, Brand-de Wilde OM, Fassbinder E, Harper RP, Lavender A, Lockwood G, Malogiannis IA, Ruths FA, Schweiger U, Shaw IA, Zarbock G, Farrell JM. Effectiveness of Predominantly Group Schema Therapy and Combined Individual and Group Schema Therapy for Borderline Personality Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Apr 1;79(4):287-299. doi: 10.1001/jamapsychiatry.2022.0010. PMID 35234828
- [Background] Bandelow B, Krause J, Wedekind D, Broocks A, Hajak G, Ruther E. Early traumatic life events, parental attitudes, family history, and birth risk factors in patients with borderline personality disorder and healthy controls. Psychiatry Res. 2005 Apr 15;134(2):169-79. doi: 10.1016/j.psychres.2003.07.008. PMID 15840418
- [Background] Brewin CR, Cloitre M, Hyland P, Shevlin M, Maercker A, Bryant RA, Humayun A, Jones LM, Kagee A, Rousseau C, Somasundaram D, Suzuki Y, Wessely S, van Ommeren M, Reed GM. A review of current evidence regarding the ICD-11 proposals for diagnosing PTSD and complex PTSD. Clin Psychol Rev. 2017 Dec;58:1-15. doi: 10.1016/j.cpr.2017.09.001. Epub 2017 Sep 6. PMID 29029837
- [Background] Cloitre M, Garvert DW, Brewin CR, Bryant RA, Maercker A. Evidence for proposed ICD-11 PTSD and complex PTSD: a latent profile analysis. Eur J Psychotraumatol. 2013 May 15;4. doi: 10.3402/ejpt.v4i0.20706. Print 2013. PMID 23687563
- [Background] Gilbar O, Hyland P, Cloitre M, Dekel R. ICD-11 complex PTSD among Israeli male perpetrators of intimate partner violence: Construct validity and risk factors. J Anxiety Disord. 2018 Mar;54:49-56. doi: 10.1016/j.janxdis.2018.01.004. Epub 2018 Jan 31. PMID 29421372
- [Background] Karatzias T, Hyland P, Bradley A, Cloitre M, Roberts NP, Bisson JI, Shevlin M. Risk factors and comorbidity of ICD-11 PTSD and complex PTSD: Findings from a trauma-exposed population based sample of adults in the United Kingdom. Depress Anxiety. 2019 Sep;36(9):887-894. doi: 10.1002/da.22934. Epub 2019 Jul 3. PMID 31268218
- [Background] Karatzias T, Shevlin M, Fyvie C, Hyland P, Efthymiadou E, Wilson D, Roberts N, Bisson JI, Brewin CR, Cloitre M. An initial psychometric assessment of an ICD-11 based measure of PTSD and complex PTSD (ICD-TQ): Evidence of construct validity. J Anxiety Disord. 2016 Dec;44:73-79. doi: 10.1016/j.janxdis.2016.10.009. Epub 2016 Oct 17. PMID 27776256
- [Background] Kilpatrick DG, Resnick HS, Milanak ME, Miller MW, Keyes KM, Friedman MJ. National estimates of exposure to traumatic events and PTSD prevalence using DSM-IV and DSM-5 criteria. J Trauma Stress. 2013 Oct;26(5):537-47. doi: 10.1002/jts.21848. PMID 24151000
- [Background] Lanius RA, Brand B, Vermetten E, Frewen PA, Spiegel D. The dissociative subtype of posttraumatic stress disorder: rationale, clinical and neurobiological evidence, and implications. Depress Anxiety. 2012 Aug;29(8):701-8. doi: 10.1002/da.21889. Epub 2012 Mar 16. PMID 22431063
- [Background] Maercker A, Brewin CR, Bryant RA, Cloitre M, Reed GM, van Ommeren M, Humayun A, Jones LM, Kagee A, Llosa AE, Rousseau C, Somasundaram DJ, Souza R, Suzuki Y, Weissbecker I, Wessely SC, First MB, Saxena S. Proposals for mental disorders specifically associated with stress in the International Classification of Diseases-11. Lancet. 2013 May 11;381(9878):1683-5. doi: 10.1016/S0140-6736(12)62191-6. Epub 2013 Apr 11. No abstract available. PMID 23583019
- [Background] Powers A, Fani N, Carter S, Cross D, Cloitre M, Bradley B. Differential predictors of DSM-5 PTSD and ICD-11 complex PTSD among African American women. Eur J Psychotraumatol. 2017 Jun 15;8(1):1338914. doi: 10.1080/20008198.2017.1338914. eCollection 2017. PMID 28649302
- [Background] Resick PA, Bovin MJ, Calloway AL, Dick AM, King MW, Mitchell KS, Suvak MK, Wells SY, Stirman SW, Wolf EJ. A critical evaluation of the complex PTSD literature: implications for DSM-5. J Trauma Stress. 2012 Jun;25(3):241-51. doi: 10.1002/jts.21699. PMID 22729974
- [Background] van der Kolk BA, Pelcovitz D, Roth S, Mandel FS, McFarlane A, Herman JL. Dissociation, somatization, and affect dysregulation: the complexity of adaptation of trauma. Am J Psychiatry. 1996 Jul;153(7 Suppl):83-93. doi: 10.1176/ajp.153.7.83. PMID 8659645